CLINICAL TRIAL: NCT07120971
Title: A Phase 0/Phase 1 Trial of Metformin for Premature Infants With Bronchopulmonary Dysplasia
Brief Title: Metformin for Premature Infants With Bronchopulmonary Dysplasia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, G. Ganesh Konduri, Professor, Division Chief of Neonatology, Medical College of Wisconsin
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: PRO55881
Record Dates: First submitted 2025-07-29; First posted 2025-08-13 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Bronchopulmonary Dysplasia (BPD)
Keywords: bronchopulmonary dysplasia; BPD; prematurity; metformin
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Phase 0 - Cohort 1 (Experimental): 5mg/kg/day in two divided doses for three days
  Interventions: Drug: Metformin (open-label)
- Phase 0 - Cohort 2 (Experimental): 10mg/kg/day in two divided doses for three days
  Interventions: Drug: Metformin (open-label)
- Phase 0 - Cohort 3 (Experimental): 20mg/kg/day in two divided doses for seven days
  Interventions: Drug: Metformin (open-label)
- Phase 0 - Cohort 4 (Experimental): 25mg/kg/day in two divided doses for 14 days
  Interventions: Drug: Metformin (open-label)
- Phase 1 - Cohort 1 Escalation (Experimental): 15mg/kg/day in a single daily dose for three days
  Interventions: Drug: Metformin (open-label)
- Phase 1 - Cohort 2 Escalation (Experimental): 25mg/kg/day in a single daily dose for three days
  Interventions: Drug: Metformin (open-label)
- Phase 1- Cohort 3 Escalation (Experimental): 10mg/kg/day in a single daily dose for three days
  Interventions: Drug: Metformin (open-label)
- Phase 1 - Cohort 4 Expansion (Experimental): 10-25mg/kg/day (dose selected from either Cohort 2 or 3)
  Interventions: Drug: Metformin (open-label)
- Phase 1 - Cohort 5 Expansion (Experimental): 10-25mg/kg/day (dose selected from either Cohort 2 or 3)
  Interventions: Drug: Metformin (open-label)

INTERVENTIONS:
Drug: Metformin (open-label) — Enteric metformin 5mg/kg/day in two divided doses will be given for three days to two subjects
  Arms: Phase 0 - Cohort 1
Drug: Metformin (open-label) — Enteric metformin 10mg/kg/day in two divided doses will be given for three days to two subjects.
  Arms: Phase 0 - Cohort 2
Drug: Metformin (open-label) — Enteric metformin 20mg/kg/day in two divided doses will be given for seven days to three subjects.
  Arms: Phase 0 - Cohort 3
Drug: Metformin (open-label) — Enteric metformin 25mg/kg/day in two divided doses will be given for 14 days to three subjects.
  Arms: Phase 0 - Cohort 4
Drug: Metformin (open-label) — Enteric metformin 15mg/kg/day in a single daily dose will be given for three days to 3-6 subjects. Depending on tolerance, the next Cohort will increase to 25mg/kg/day (Cohort 2) or decrease to 10mg/kg/day (Cohort 3)
  Arms: Phase 1 - Cohort 1 Escalation
Drug: Metformin (open-label) — Enteric metformin 25mg/kg/day in a single daily dose will be given for three days to 3-6 subjects. Depending on tolerance, either 25mg/kg/day or 15mg/kg/day will be dose selected for the next Cohort (Cohort 4)
  Arms: Phase 1 - Cohort 2 Escalation
Drug: Metformin (open-label) — Enteric metformin 10mg/kg/day in a single daily dose will be given for three days to 3-6 subjects. Depending on tolerance, either 10mg/kg/day dose selected for the next Cohort (Cohort 4) or the study will be stopped due to excessive toxicity.
  Arms: Phase 1- Cohort 3 Escalation
Drug: Metformin (open-label) — The dose for this cohort will be selected from either Cohort 2 or 3 based on tolerance. Enteric metformin 10-25mg/kg/day in a single daily dose will be given for seven days to 6 subjects.
  Arms: Phase 1 - Cohort 4 Expansion
Drug: Metformin (open-label) — The dose for this cohort will be the same as Cohort 4. Enteric metformin 10-25mg/kg/day in a single daily dose will be given for 14 days to 6 subjects.
  Arms: Phase 1 - Cohort 5 Expansion

SUMMARY:
The overall objective of this study is to investigate the role of metformin in decreasing lung injury and promoting lung growth in premature infants. There are two phases to this pilot study. For Phase 0, the goal is to investigate the safety and tolerance of oral metformin in premature who have been diagnosed with bronchopulmonary dysplasia (BPD) at 36-44 weeks gestation. For Phase 1, the goal is to investigate metformin safety and tolerance in extremely premature infants who are 7-30 days old who have an increased risk of BPD. The main questions it aims to answer are:

* how well do older premature infants tolerate metformin?
* how well do younger premature infants tolerate metformin?

DETAILED DESCRIPTION:
In Phase 0, there are four groups with different doses of metformin, starting at 5mg/kg/day to a maximum of 25mg/kg/day. Participants will take oral metformin twice a day for 3, 7 or 14 days, depending on which group they are in. In Phase 1, there are four groups with different doses of metformin, starting at 15mg/kg/day to a maximum of 25mg/kg/day. Participants will take oral metformin once a day for 3, 7, or 14 days, depending on what group they are in.

ELIGIBILITY:
Inclusion Criteria Phase 0:

* Birth gestational age of < 29 weeks AND
* Postnatal age between 8 and 22 weeks AND
* Diagnosed with BPD at 36 weeks postnatal age

Inclusion Criteria Phase 1:

* Birth gestational age of < 29 weeks, AND
* Requiring mechanical ventilation or positive pressure support at 7 days postnatal age, AND
* Postnatal age between 7 and 30 days

Exclusion Criteria:

* Persistent hypoglycemia
* Lactic acidosis
* Feeding intolerance
* Renal or hepatic dysfunction
* Active infection
* Congenital anomalies that preclude feedings
* Infants whose parents have chosen palliative care

Ages: 7 Days to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who tolerate metformin | 14 days after administration of the first dose of metformin
  Number of subjects who receive enteral doses of metformin and complete the study days without an adverse event while continuing enteral feedings
Number of participants with treatment-related adverse events | 14 days after administration of the first dose of metformin
  Number of participants who develop hypoglycemia defined as blood glucose value <50
Number of participants with treatment-related metabolic acidosis | 14 days after administration of the first dose of metformin
  Number of subjects who develop lactic acid levels > 5mmol/L
Number of subjects with treatment-related feeding problems | 14 days after administration of the first dose of metformin
  Number of subjects who require a decrease in enteral feeding volume by >50% from baseline
Number of subjects who require dose adjustments of metformin | 14 days after administration of the first dose of metformin
  Number of subjects who need decreases in dose or discontinuation of metformin due to hepatic or renal dysfunction
Number of subjects with respiratory deterioration | 14 days after administration of the first dose of metformin
  Number of subjects who develop pneumonia and increases in oxygen concentration and ventilator support during the study
Number of subjects who complete pharmacokinetic evaluation of metformin | 14 days after administration of the first dose of metformin
  Number of subjects who have at least one metformin concentration in blood measured at 1, 4 and 12 hours after an enteric dose
Pharmacokinetic analysis of metformin | 14 days after administration of the first dose of metformin
  Area under the curve of Plasma Concentration Versus Time (AUC) of metformin over a time frame of 1, 4 and 12 hours after an enteric dose of metformin.
Number of subjects who complete the treatment protocol | 14 days after administration of the first dose of metformin
  Number of subjects who complete the study doses of enteric metformin

SECONDARY OUTCOMES:
Incidence of bronchopulmonary dysplasia | 14 days after administration of the first dose of metformin
  Number of subjects who are diagnosed with bronchopulmonary dysplasia
Incidence of necrotizing enterocolitis | 14 days after administration of the first dose of metformin
  Number of subjects who are diagnosed with necrotizing enterocolitis
Incidence of retinopathy of prematurity | 14 days after administration of the first dose of metformin
  Number of subjects who are diagnosed with retinopathy of prematurity
Incidence of intraventricular hemorrhage | 14 days after administration of the first dose of metformin
  Number of subjects who are diagnosed with intraventricular hemorrhage
Incidence of patent ductus arteriosus | 14 days after administration of the first dose of metformin
  Number of subjects who are diagnosed with patent ductus arteriosus

CONTACTS AND LOCATIONS:
Overall Officials: G. Ganesh Konduri, MD, MS, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
Since this is a small phase 0 and phase 1 study with enrollment of 4-30 infants from one site only in a short time frame, we are concerned about potential for unmasking the identification of individual identification from the sharing of individual patient data.

REFERENCES:
- [Background] Rana U, Joshi C, Whitney E, Afolayan A, Dowell J, Teng RJ, Konduri GG. Decreased Liver Kinase B1 Expression and Impaired Angiogenesis in a Murine Model of Bronchopulmonary Dysplasia. Am J Respir Cell Mol Biol. 2024 Oct;71(4):481-494. doi: 10.1165/rcmb.2024-0037OC. PMID 38869353
- [Background] Alemon-Medina R, Altamirano-Bustamante N, Lugo-Goytia G, Garcia-Alvarez R, Rivera-Espinosa L, Torres-Espindola LM, Chavez-Pacheco JL, Juarez-Olguin H, Gomez-Garduno J, Flores-Perez C, Fernandez-Perez PG. Comparative Bioavailability and Pharmacokinetics Between the Solid Form of Metformin vs a Novel Liquid Extemporaneous Formulation in Children. Dose Response. 2021 Sep 27;19(3):15593258211033140. doi: 10.1177/15593258211033140. eCollection 2021 Jul-Sep. PMID 34602916
- [Background] Kirkpatrick EC, Mitchell ME, Thilly WG, Cava J, Tomita-Mitchell A, Gostjeva EV. Use of Metformin in Pulmonary Vein Stenosis after TAPVR Repair. Glob Pediatr Health. 2020 Sep 25;7:2333794X20958924. doi: 10.1177/2333794X20958924. eCollection 2020. No abstract available. PMID 33029553
- [Background] Ayoub R, Ruddy RM, Cox E, Oyefiade A, Derkach D, Laughlin S, Ades-Aron B, Shirzadi Z, Fieremans E, MacIntosh BJ, de Medeiros CB, Skocic J, Bouffet E, Miller FD, Morshead CM, Mabbott DJ. Assessment of cognitive and neural recovery in survivors of pediatric brain tumors in a pilot clinical trial using metformin. Nat Med. 2020 Aug;26(8):1285-1294. doi: 10.1038/s41591-020-0985-2. Epub 2020 Jul 27. PMID 32719487
- [Background] Biag HMB, Potter LA, Wilkins V, Afzal S, Rosvall A, Salcedo-Arellano MJ, Rajaratnam A, Manzano-Nunez R, Schneider A, Tassone F, Rivera SM, Hagerman RJ. Metformin treatment in young children with fragile X syndrome. Mol Genet Genomic Med. 2019 Nov;7(11):e956. doi: 10.1002/mgg3.956. Epub 2019 Sep 14. PMID 31520524
- [Background] Brittain EL, Niswender K, Agrawal V, Chen X, Fan R, Pugh ME, Rice TW, Robbins IM, Song H, Thompson C, Ye F, Yu C, Zhu H, West J, Newman JH, Hemnes AR. Mechanistic Phase II Clinical Trial of Metformin in Pulmonary Arterial Hypertension. J Am Heart Assoc. 2020 Nov 17;9(22):e018349. doi: 10.1161/JAHA.120.018349. Epub 2020 Nov 10. PMID 33167773
- [Background] Liao S, Li D, Hui Z, McLachlan CS, Zhang Y. Metformin added to bosentan therapy in patients with pulmonary arterial hypertension associated with congenital heart defects: a pilot study. ERJ Open Res. 2018 Aug 22;4(3):00060-2018. doi: 10.1183/23120541.00060-2018. eCollection 2018 Jul. PMID 30151369
- [Background] Wang X, Liu Y, Han D, Zhong J, Yang C, Chen X. Dose-dependent immunomodulatory effects of metformin on human neonatal monocyte-derived macrophages. Cell Immunol. 2022 Jul;377:104557. doi: 10.1016/j.cellimm.2022.104557. Epub 2022 Jun 3. PMID 35679651
- [Background] Jing Y, Wu F, Li D, Yang L, Li Q, Li R. Metformin improves obesity-associated inflammation by altering macrophages polarization. Mol Cell Endocrinol. 2018 Feb 5;461:256-264. doi: 10.1016/j.mce.2017.09.025. Epub 2017 Sep 18. PMID 28935544
- [Background] Howie SR. Blood sample volumes in child health research: review of safe limits. Bull World Health Organ. 2011 Jan 1;89(1):46-53. doi: 10.2471/BLT.10.080010. Epub 2010 Sep 10. PMID 21346890
- [Background] Autmizguine J, Benjamin DK Jr, Smith PB, Sampson M, Ovetchkine P, Cohen-Wolkowiez M, Watt KM. Pharmacokinetic studies in infants using minimal-risk study designs. Curr Clin Pharmacol. 2014;9(4):350-8. doi: 10.2174/1574884709666140520153308. PMID 24844642
- [Background] General clinical pharmacology considerations for neonatal studies for drugs and biological products- Guidance for industry. Food and Drug Administration. Clinical Pharmacology July 2022
- [Background] See KC. Metformin-associated lactic acidosis: A mini review of pathophysiology, diagnosis and management in critically ill patients. World J Diabetes. 2024 Jun 15;15(6):1178-1186. doi: 10.4239/wjd.v15.i6.1178. PMID 38983827
- [Background] Le Tourneau C, Lee JJ, Siu LL. Dose escalation methods in phase I cancer clinical trials. J Natl Cancer Inst. 2009 May 20;101(10):708-20. doi: 10.1093/jnci/djp079. Epub 2009 May 12. PMID 19436029
- [Background] DeFronzo R, Fleming GA, Chen K, Bicsak TA. Metformin-associated lactic acidosis: Current perspectives on causes and risk. Metabolism. 2016 Feb;65(2):20-9. doi: 10.1016/j.metabol.2015.10.014. Epub 2015 Oct 9. PMID 26773926
- [Background] Hutchinson AM, Pais R, Endginton AN, Pilon B, MacDonald JM, MacDonald ME, Lewis T, Offringa M, Kalish BT. Safety and feasibility trial protocol of metformin in infants after perinatal brain injury. BMJ Paediatr Open. 2025 Aug 24;9(1):e002784. doi: 10.1136/bmjpo-2024-002784. PMID 40850908
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Abman SH, Bancalari E, Jobe A. The Evolution of Bronchopulmonary Dysplasia after 50 Years. Am J Respir Crit Care Med. 2017 Feb 15;195(4):421-424. doi: 10.1164/rccm.201611-2386ED. No abstract available. PMID 28199157
- [Background] Hardie DG, Ross FA, Hawley SA. AMPK: a nutrient and energy sensor that maintains energy homeostasis. Nat Rev Mol Cell Biol. 2012 Mar 22;13(4):251-62. doi: 10.1038/nrm3311. PMID 22436748
- [Background] Park SI, Lee H, Oh J, Lim KS, Jang IJ, Kim JA, Jung JH, Yu KS. A fixed-dose combination tablet of gemigliptin and metformin sustained release has comparable pharmacodynamic, pharmacokinetic, and tolerability profiles to separate tablets in healthy subjects. Drug Des Devel Ther. 2015 Feb 4;9:729-36. doi: 10.2147/DDDT.S75980. eCollection 2015. PMID 25678778
- [Background] Kuhlmann I, Noddebo Nyrup A, Bjerregaard Stage T, Hougaard Christensen MM, Korshoj Bergmann T, Damkier P, Nielsen F, Hojlund K, Brosen K. Oral and intravenous pharmacokinetics of metformin with and without oral codeine intake in healthy subjects: A cross-over study. Clin Transl Sci. 2021 Nov;14(6):2408-2419. doi: 10.1111/cts.13107. Epub 2021 Aug 12. PMID 34268884
- [Background] Yadav A, Rana U, Michalkiewicz T, Teng RJ, Konduri GG. Decreased AMP-activated protein kinase (AMPK) function and protective effect of metformin in neonatal rat pups exposed to hyperoxia lung injury. Physiol Rep. 2020 Sep;8(18):e14587. doi: 10.14814/phy2.14587. PMID 32959498
- [Background] Ratner V, Starkov A, Matsiukevich D, Polin RA, Ten VS. Mitochondrial dysfunction contributes to alveolar developmental arrest in hyperoxia-exposed mice. Am J Respir Cell Mol Biol. 2009 May;40(5):511-8. doi: 10.1165/rcmb.2008-0341RC. Epub 2009 Jan 23. PMID 19168698

DOCUMENTS (1):
  • Informed Consent Form (2025-08-25): https://cdn.clinicaltrials.gov/large-docs/71/NCT07120971/ICF_000.pdf